CLINICAL TRIAL: NCT06664281
Title: Effects of Sprint Interval Training Combined with Remote Ischemic Preconditioning on Vascular Function in Young Women with Masked Obesity
Brief Title: Effects of SIT Combined with Remote Ischemic Preconditioning on Vascular Function in Young Women with Masked Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESITCRIPVFYWMO
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Vascular Function
Keywords: Sprint Interval Training; Masked Obesity; Young Women; Ischemic Preconditioning; Vascular Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- sprint interval training group (Active Comparator)
  Interventions: Behavioral: SIT
- sprint interval training combined with remote ischemic preconditioning group (Active Comparator)
  Interventions: Behavioral: SIT combined RIPC
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: SIT — sprint interval training
  Arms: sprint interval training group
Behavioral: SIT combined RIPC — sprint interval training combined with remote ischemic preconditioning
  Arms: sprint interval training combined with remote ischemic preconditioning group

SUMMARY:
Comparison of the effects of combined Sprint Interval Training (SIT) with Remote Ischemic Preconditioning (RIPC) and SIT on vascular function in young women with masked obesity.

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 3 arms (control group, SIT group and SIT with RIPC group), in which a pre-treatment-posttest design has been used.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 and 30 years;
* BMI within the normal range (18.5～24.9 kg/m²), BF% > 30%;
* Participants with no clinically diagnosed contraindications for exercise, in good health, and not engaged in regular exercise, as determined by the health and physical activity questionnaire (based on the American College of Sports Medicine's guidelines for exercise testing and prescription).

Exclusion Criteria:

* History of cardiovascular diseases, including coronary heart disease, stroke, or peripheral arterial disease diagnosed through vascular imaging techniques;
* Currently participating in other intervention studies, including dietary, nutritional, or psychological education programs;
* Those with regular professional training;
* Musculoskeletal disorders that make long-term exercise interventions unsuitable.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Intima-Media Thickness (IMT) | 8 weeks
  Changes in Intima media thickness before and after intervention.
Flow-Mediated Dilation (FMD) | 8 weeks
  Changes in Flow-mediated dilation before and after Intervention. Brachial artery flow-mediated dilation (FMD) was measured by the UNEXEF high-resolution ultrasound vascular endothelial function analyzer.

SECONDARY OUTCOMES:
Body Composition Indicator | 8 weeks
  Changes in Body composition indicators before and after Intervention. Including body fat percentage (BF%).
Human Morphometric i Indicators | 8 weeks
  Changes in Human morphometric indicators before and after Intervention. Including height, weight, waist circumference, hip circumference, and body mass index (BMI). BMI was calculated based on the measured height and weight using the formula: BMI = weight/height² (kg/m²).
Blood Pressure (BP) | 8 weeks
  Changes in blood pressure before and after intervention. Including systolic and diastolic blood pressure.
Nitric Oxide (NO) | 8 weeks
  Changes in concentration of nitric oxide before and after Intervention.
Maximum Oxygen Uptake (VO2max) | 8 weeks
  Changes in maximum oxygen uptake before and after Intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China

REFERENCES:
- [Derived] Ji Y, Yang L, Zhang P. Effects of sprint interval training combined with remote ischaemic preconditioning on vascular function in young women with masked obesity. Eur J Appl Physiol. 2025 Sep 22. doi: 10.1007/s00421-025-05970-4. Online ahead of print. PMID 40982049